CLINICAL TRIAL: NCT00251615
Title: Calcium Channel Splice Variant Expression in Cardiovascular Disease and Aging
Status: Completed | Type: Observational
Sponsor: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: AG0058
Record Dates: First submitted 2005-11-08; First posted 2005-11-10 (Estimated); Last update posted 2012-08-06 (Estimated); Status verified 2012-08

CONDITIONS: Atherosclerosis
Keywords: vascular surgery; vascular aging; arterial aging; surgical tissue; Aging
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Vascular tissue obtained from the surgical site that would have otherwise been discarded and Blood Serum

SUMMARY:
The purpose of this study is to learn what changes in blood vessel contraction may occur as a result of a disease of the vessel that requires surgery. The study will examine the calcium channels present in the vessels being operated on, and the genes that may alter blood vessel function. Possible variation in these genes may change the kind of calcium channels present in blood vessels.

DETAILED DESCRIPTION:
The goal of this study is to learn more about how blood vessels function and the mechanism that causes them to contract. The study will investigate the natural history of diseased blood vessel tissue and the calcium channels in the muscle part of the blood vessel. The study will also examine how genetics influences cardiovascular disease and its causes and treatments.

Patients scheduled for vascular surgery will be approached to participate in this study. During surgery, tissue fragments of diseased and marginal tissue will be obtained. A blood sample will be obtained at either the time of surgery or consent and genomic DNA will be extracted.

ELIGIBILITY:
Inclusion Criteria:

* Ages 21 and older
* Scheduled for vascular surgery

Exclusion Criteria:

* Unwillingness to be subjected to diagnostic and/or therapeutic procedures that are deemed not necessary for clinical management
* Volunteers deemed too fragile to participate in the study by the principal investigator (PI) or the attending physician
* Inability to obtain informed consent from either the volunteer or the responsible party (durable power of attorney [DPA]) for the volunteer, with the volunteer's assent

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for vascular surgery
Sampling Method: Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2012-08; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samer Najjar, MD, Principal Investigator — National Institute on Aging (NIA)
Locations (1):
- National Institute on Aging, Harbor Hospital, Baltimore, Maryland, United States

REFERENCES:
- [Background] Harry JB, Kobrinsky E, Abernethy DR, Soldatov NM. New short splice variants of the human cardiac Cavbeta2 subunit: redefining the major functional motifs implemented in modulation of the Cav1.2 channel. J Biol Chem. 2004 Nov 5;279(45):46367-72. doi: 10.1074/jbc.M409523200. Epub 2004 Aug 31. PMID 15339916
- [Background] Kobrinsky E, Tiwari S, Maltsev VA, Harry JB, Lakatta E, Abernethy DR, Soldatov NM. Differential role of the alpha1C subunit tails in regulation of the Cav1.2 channel by membrane potential, beta subunits, and Ca2+ ions. J Biol Chem. 2005 Apr 1;280(13):12474-85. doi: 10.1074/jbc.M412140200. Epub 2005 Jan 25. PMID 15671035
- [Background] Abernethy DR, Soldatov NM. Structure-functional diversity of human L-type Ca2+ channel: perspectives for new pharmacological targets. J Pharmacol Exp Ther. 2002 Mar;300(3):724-8. doi: 10.1124/jpet.300.3.724. PMID 11861774